CLINICAL TRIAL: NCT07171060
Title: Laplace Outside the US (OUS) Early Feasibility Study (EFS) Canada
Brief Title: Laplace Early Feasibility Study - Canada
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laplace Interventional, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN-003
Record Dates: First submitted 2025-08-28; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Tricuspid Valve Replacement (Experimental): Transcatheter Tricuspid Valve Replacement (TTVR) System for the treatment of severe, symptomatic tricuspid regurgitation
  Interventions: Device: Laplace TTVR System

INTERVENTIONS:
Device: Laplace TTVR System — Transcatheter Tricuspid Valve Replacement (TTVR) System for the treatment of severe, symptomatic tricuspid regurgitation

SUMMARY:
The objective of the study is to assess the safety and technical feasibility of the Laplace Transcatheter Tricuspid Valve Replacement (TTVR) System

DETAILED DESCRIPTION:
Early Feasibility (EFS), prospective, single-arm, multi-center study to evaluate safety and technical feasibility of the Laplace TTVR System in the treatment of severe, symptomatic tricuspid regurgitation patients.

ELIGIBILITY:
Inclusion Criteria:

1. 60 - 90 years of age at the time of the study procedure
2. Symptomatic tricuspid regurgitation despite being adequately treated with optimal medical therapy by the Local Heart Team for at least 30 days prior to the time of study consent.
3. Severe, massive or torrential tricuspid regurgitation determined by qualifying transthoracic echocardiogram (TTE) and/or transesophageal echocardiogram (TEE) using the 5-grade classification.
4. Candidate felt suitable for transcatheter tricuspid valve replacement as determined by the local heart team and confirmed by the patient selection committee. For patients with pre-existing trans-tricuspid pacemaker or ICD leads, the local heart team shall include an electrophysiologist.
5. Anatomically suitable for the Laplace TTVR system including trans-jugular access 6 Subject or legally authorized representative has provided informed consent and agrees to return for all required post-procedure follow-up visits

Exclusion Criteria:

1. Estimated life expectancy of less than 12 months
2. Systolic pulmonary artery pressure > 65mmHg per TTE.
3. PVR >5 Wood units
4. Acutely decompensated defined as hypotension with SBP <90 mmHg, use of hemodynamic support devices or inotropes within the last 30 days
5. Severe COPD dependent on home oxygen or chronic home oxygen use
6. Echocardiographic evidence of severe right ventricular dysfunction
7. Severe aortic, mitral and/or pulmonic valve stenosis and/or regurgitation requiring treatment
8. New or untreated right heart chamber or/and superior vena cava intracardiac mass, thrombus, or vegetation
9. Presence of significant congenital heart disease including but not limited to hemodynamically significant atrial septal defect, RV dysplasia, and arrhythmogenic RV.
10. Untreatable hypersensitivity or contraindication to any of the following: Aspirin, and Clopidogrel or Ticlopidine, Heparin, and Bivalirudin, Warfarin, or DOAC, Nitinol Alloys. Severe renal insufficiency defined as eGFR <25 mL/min or requiring chronic renal replacement therapy at the time of screening committee review.

12. Current history (within last 5 years) of illicit drug use. 13. Any percutaneous cardiovascular intervention, cardiovascular surgery, or carotid surgery, within last 30 days. Implant or revision of any rhythm management device (CRT or CRT-D) or implantable cardioverter-defibrillator or leadless pacemaker within 90 days prior to the study procedure 14. Need for emergent, urgent or planned surgery or intervention within 30 days following the study procedure. Planned or scheduled cardiac surgery within next 12 months. 15. Stroke or other major cerebrovascular event within 90-days prior to index procedure 16. Untreated clinically significant coronary artery disease requiring revascularization, recent (within last 30 days) acute coronary syndrome or myocardial infarction. 17. Active or recent GI bleed within 30 days prior to study procedure or patients Contraindicated for oral anticoagulation therapy 18. Bleeding disorders including thrombocytopenia or platelet count <70,000 mm 3 or thrombocytosis (platelet count >700,000 /mm 3

* Transfusion dependent chronic anemia with Hb <9/dL
* Current or planned pregnancy within next 12 months for women of childbearing potential
* Active or recent endocarditis within last 90 days or, sepsis/ other systemic infection requiring oral or intravenous antibiotics within last 30 days
* Prior tricuspid repair or tricuspid replacement or other device that would interfere with successful deployment or functioning of Laplace tricuspid valve.
* Participation in another pre-market investigational device study or investigational drug study for a cardiac related drug
* Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements. Any patient considered to be vulnerable.
* Left ventricular ejection fraction (LVEF) < 30%
* Deep vein thrombosis or pulmonary embolism within last 6 months
* Child-Pugh C cirrhosis.
* Contraindication or inability to complete TEE

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Technical success | During procedure
  Successful valve implantation

SECONDARY OUTCOMES:
Procedural success | During procedure
  Tricuspid regurgitation of moderate or less
Device success | 30-days post-procedure
  Freedom from reintervention due to device related complications

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Research Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No